CLINICAL TRIAL: NCT03983889
Title: The Effect and Safety of Different Sedation Strategies for Diagnostic Bronchoscopy
Brief Title: Sedation Strategies for Diagnostic Bronchoscopy 2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Changhai Hospital (Other)
Collaborators: Shanghai Zhongshan Hospital (Other); Ruijin Hospital (Other); Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, Jia-feng Wang, Clinical Professor, Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SED-DFB2
Record Dates: First submitted 2019-06-10; First posted 2019-06-12 (Actual); Last update posted 2019-06-14 (Actual); Status verified 2019-06

CONDITIONS: Bronchoscopy; Sedation
MeSH Terms: interventions — Midazolam; Fentanyl; Dexmedetomidine; Remifentanil; Propofol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- F (Experimental): Sedated with intravenous midazolam (0.03mg/kg) and fentanyl (1μg/kg) for induction and maintenance
  Interventions: Drug: Midazolam; Drug: Fentanyl
- DR (Experimental): Sedated with intravenous midazolam (0.03mg/kg), dexmedetomidine (0.5-1μg/kg for induction+0.5-0.7μg/kg/h for maintenance) and remifentanil (plasma concentration 2.0-2.5ng/ml) for induction and maintenance
  Interventions: Drug: Midazolam; Drug: Dexmedetomidine; Drug: Remifentanil
- DF (Experimental): Sedated with intravenous midazolam (0.03mg/kg), dexmedetomidine (0.5-1μg/kg for induction+0.5-0.7μg/kg/h for maintenance) and fentanyl (1μg/kg) for induction and maintenance
  Interventions: Drug: Midazolam; Drug: Fentanyl; Drug: Dexmedetomidine
- PR (Experimental): Sedated with intravenous midazolam (0.03mg/kg), propofol (plasma concentration 1.0-2.0ng/ml) and remifentanil (plasma concentration 2.0-2.5ng/ml) for induction and maintenance
  Interventions: Drug: Midazolam; Drug: Remifentanil; Drug: Propofol

INTERVENTIONS:
Drug: Midazolam — Midazolam is used as a common medication for sedation in all groups.
Drug: Fentanyl — Fentanyl is another opioid drug used for analgesia to prevent bronchoscopy induced cough.
  Arms: DF; F
Drug: Dexmedetomidine — Dexmedetomidine is used for sedation in bronchoscopy with less impact on respiration.
  Arms: DF; DR
Drug: Remifentanil — Remifentanil is used for analgesia to prevent bronchoscopy induced cough.
  Arms: DR; PR
Drug: Propofol — Propofol is used for sedation with high efficacy but more side effect on respiration than dexmedetomidine.
  Arms: PR

SUMMARY:
Diagnostic bronchoscopy is an invasive procedure performed to diagnose respiratory diseases. But pain has been complained by most of the patients receiving such procedures. Sedation or anesthesia was required by both of the patients and bronchoscopists. Unfortunately, no consensus has been made upon the sedation strategies. Multiple sedation approaches have been applied, such as midazolam and fentanyl, remifentanil and propofol, dexmedetomidine and propofol. The present study was designed to compare these protocols in sedation for diagnostic bronchoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for flexible diagnostic bronchoscopy
* Adult patients aged 18 to 65 years
* American Society of Anesthesiologists (ASA) Physical Status Classification I-II
* BMI 18.5-25kg/m2
* Subjects provide informed consent

Exclusion Criteria:

* Severe airway obstruction
* Coagulation disorder
* Repeat bronchoscopy (more than 3 times)
* Severe liver and renal dysfunction
* Cardiovascular and cerebrovascular diseases
* Pregnancy
* Chronic opioid user
* Drug abusers or addicts

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-06-17 (Estimated); Primary Completion 2019-11-30 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Cough score | From the completion of local anesthesia with lidocaine to the completion of bronchoscopy procedure, assessed up to 2 hours
  Cough score across the procedure will be classified into 4 degree (1-4) as follows. 1 = none, 2 = one gag or cough only, 3 = >1 gag or cough, but acceptable conditions, 4 = unacceptable conditions

SECONDARY OUTCOMES:
Body movement | From the completion of local anesthesia with lidocaine to the completion of bronchoscopy procedure, assessed up to 2 hours
  The numbers of the times of any body movement across the procedure
Satisfaction score of the patients and bronchoscopists | Across the procedure, assessed up to 2 hours
  Satisfaction score of the patients and bronchoscopists regarding to the sedation quality measured by a 0-100 visual analogue scale (VAS). 100 refers to the highest satisfaction degree while 0 refers to the worst satisfaction degree. The scale score was determined by the subjective determination of the satisfaction on the sedation quality.
Amount of the rescue use of propofol | After sedation induction, assessed up to 2 hours
  The total amount of propofol used as a rescue therapy when the sedation is not deep enough as assessed by the anesthesiologists.
Recovery time | After termination of the sedation medication, assessed up to 2 hours
  Duration of the recovery from sedation
Prevalence of the side effects of respiratory and circulatory system | Across the sedation duration, assessed up to 2 hours
  The number of the side effects in respiratory and circulatory system during the procedure, including hypertension, hypotension, tachycardia, bradycardia, hypoxia and larynx spasm.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Anesthesiology, Changhai Hospital, Shanghai, Shanghai Municipality, China